CLINICAL TRIAL: NCT06699849
Title: A Phase 2, Multicenter, Randomized, Multiple-Dose, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of CSL889 in Adults and Adolescents With Sickle Cell Disease During Vaso-Occlusive Crisis
Brief Title: Safety, Efficacy, and Pharmacokinetics of CSL889 in Adults and Adolescents With Sickle Cell Disease During Vaso-Occlusive Crisis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL889_2001; 2024-513440-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease Vaso-occlusive Crisis
Keywords: Sickle cell disease; Acute kidney injury; Pharmacokinetics; Acute chest syndrome; Vaso-occlusive crisis; Hemopexin
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Kidney Injury; Acute Chest Syndrome; Vaso-Occlusive Crises | interventions — Hemopexin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CSL889 Regimen 1 (Experimental): Participants in this arm will receive CSL889 as per regimen 1.
  Interventions: Biological: CSL889
- CSL889 Regimen 2 (Experimental): Participants in this arm will receive CSL889 as per regimen 2.
  Interventions: Biological: CSL889
- Placebo (Placebo Comparator): Participants in this arm will receive placebo matching to CSL889 regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CSL889 — CSL889 is a solution for infusion to be administered by the IV route.
  Other Names: Hemopexin, human
  Arms: CSL889 Regimen 1; CSL889 Regimen 2
Drug: Placebo — Volume and regimen matched to CSL889 will be administered.
  Arms: Placebo

SUMMARY:
This is a phase 2, randomized, multiple-dose, placebo-controlled study designed to evaluate the safety, efficacy, and pharmacokinetics (PK) of CSL889 (human hemopexin) when given intravenously (IV) to adults and adolescents with sickle cell disease (SCD) experiencing vaso-occlusive crises (VOC). The main objectives of the study are to evaluate the safety and tolerability of CSL889 in study participants, and to assess how CSL889 affects the time it takes for VOC to resolve in participants with SCD.

ELIGIBILITY:
Inclusion Criteria:

* At the time of informed consent:

  * 18 years of age (adults); or
  * 12 to less than (<) 18 years of age (adolescents, where approved and when enrollment for adolescents has been opened by the sponsor, with the endorsement of the Independent Data Monitoring Committee [IDMC])
* Diagnosed with SCD (any genotype).
* Presented at the study site with a new acute VOC necessitating treatment with parenteral opioids.

Exclusion Criteria:

* VOC pain onset greater than (>) 72 hours before administration of first parenteral opioid.
* Must not have a history of > 5 VOCs requiring hospital admission in the past 6 months; or signs and / or symptoms of ACS; or new neurological symptoms suggestive of acute stroke or transient ischemic attack; or any stage (acute kidney injury) AKI; or been discharged from inpatient hospital admission for VOC or other vaso-occlusive event within 14 days before the current presentation.
* Serum hemoglobin < 6 g/dL, serum ferritin ≥ 2000 ng/mL, receiving an approved medication for SCD that has not been on a stable, well-tolerated regimen, currently taking methadone or buprenorphine.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-08-07 (Estimated); Study Completion 2027-08-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to Day 28 (End of study [EOS] Visit)
Percentage of participants with TEAEs | Up to Day 28 (EOS Visit)
Number of participants with detectable treatment emergent (TE) anti-CSL889 antibodies | Up to Day 28 (EOS Visit)
Percentage of participants with detectable TE anti-CSL889 antibodies | Up to Day 28 (EOS Visit)
Time to resolution of VOC (time to discontinuation of parenteral opioids) | Up to Day 28 (EOS Visit)

SECONDARY OUTCOMES:
Hospital admission rate | Up to Day 28 (EOS Visit)
  Hospital admission rate in participants with SCD presenting with VOC who received greater than or equal to (≥) 1 dose of CSL889 in the acute care setting.
Length of hospital stay (If hospitalized) | Up to Day 28 (EOS Visit)
Percentage of participants experiencing acute chest syndrome (ACS), acute kidney injury (AKI), or stroke | From the start of investigational product (IP) administration up to Day 8
Length of acute care stay | Up to Day 28 (EOS Visit)
Total Length of acute care and hospital stay | Up to Day 28 (EOS Visit)
Re-presentation rate to an acute care facility for VOC or ACS after discharge | From discharge up to Day 28
Hospital admission rate for VOC or ACS after discharge | From discharge up to Day 28
Opioid consumption | From the time of enrollment to discharge (up to Day 28 [EOS Visit])
  Opioid consumption will be measured in morphine milligram equivalent units.
Number of participants with ≥ 30% pain reduction by Numeric Rating Scale (NRS) score | Within 4 hours after the start of CSL889 infusion
  The NRS for pain is a validated self-reported 11-point pain severity scale (where 0 means no pain and 10 means the most or worst possible pain) that can be used in adults, adolescents, and children ≥ 8 years of age with SCD.
Percentage of participants with ≥ 30% pain reduction by NRS score | Within 4 hours after the start of CSL889 infusion
  The NRS for pain is a validated self-reported 11-point pain severity scale (where 0 means no pain and 10 means the most or worst possible pain) that can be used in adults, adolescents, and children ≥ 8 years of age with SCD.
Maximum observed concentration (Cmax) after Doses 1 and 3 of CSL889 | Before dosing, and up to 12 hours after Doses 1 and 3
Area under the concentration (AUCtau) after Doses 1 and 3 of CSL889 | Before dosing, and up to 12 hours after Doses 1 and 3
Time of maximum concentration (Tmax) after Doses 1 and 3 of CSL889 | Before dosing, and up to 12 hours after Doses 1 and 3
Trough concentration (Ctrough) after each dose of CSL889 | Up to Day 5
Accumulation ratio (AR) for AUCtau of CSL889 (the ratio between the AUCtau of Doses 3 and 1) | Before dosing and at up to 12 hours after Doses 1 and 3
AR for Cmax of CSL889 (the ratio between the Cmax of Doses 3 and 1) | Before dosing and at up to 12 hours after Doses 1 and 3
AR for Ctrough of CSL889 (the ratio between the Ctrough of the last dose and Dose 1) | Before dosing and after Dose 1 and the last dose
Cmax after each dose in Sparse PK subset of CSL889 | Up to Day 5
  Sparse PK blood sampling will be performed in remainder of participants who are not in the Adult or Adolescent PK Subsets.
Ctrough after each dose in Sparse PK subset of CSL889 | Up to Day 5
  Sparse PK blood sampling will be performed in remainder of participants who are not in the Adult or Adolescent PK Subsets.
AR for Cmax in Sparse PK subset of CSL889 | Up to Day 5
  Sparse PK blood sampling will be performed in remainder of participants who are not in the Adult or Adolescent PK Subsets.
AR for Ctrough in Sparse PK subset of CSL889 | Up to Day 5
  Sparse PK blood sampling will be performed in remainder of participants who are not in the Adult or Adolescent PK Subsets.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (12):
- United States (9):
  - University of California Irvine, Orange, California
  - Golisano Children's Hospital, Fort Myers, Florida
  - The Foundation for Sickle Cell Disease, Hollywood, Florida
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mount Sinai Medical Center, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
- Turkey (Türkiye) (3):
  - Hacettepe Universitesi, Ankara
  - Istanbul Universitesi, Istanbul
  - Özel Acibadem Adana Hastanesi, Seyhan

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (i.e. FDA, EMA) is complete and the primary publication is available
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.